CLINICAL TRIAL: NCT05830357
Title: Prevalence and Risk Factors of Helicobacter Pylori Infection in Children and Young Adults in Sohag Governorate
Brief Title: Prevalence and Risk Factors of Helicobacter Pylori Infection in Children and Young Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maha Ayman Thabet, demonstrator at family medicine department, Sohag University
Other Study IDs: Soh-Med-23-04-15MS
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; dyspepsia; children; young adults; prevalence; peptic ulcer; risk factors
MeSH Terms: conditions — Dyspepsia; Peptic Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — stool specimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Helicobacter pylori is a gram-negative bacterium that resides in the stomach and can cause inflammation leading to long-term effects, such as gastric ulcers, cancer, and lymphoma of the stomach mucosal linings Previous research and analysis of H. pylori prevalence in populations have examined common risk factors that increase the likelihood of acquiring the bacteria. Some of the most commonly identified risk factors across various studies in different geographic populations are larger family size, less education, lower socioeconomic status, less frequent hygiene practices, and lower sanitation with specific emphasis on sources of water and defecation.

aim of the work: Studying prevalence of Helicobacter Pylori infection and its related risk factors in children and young adults in Sohag governorate.

ELIGIBILITY:
Inclusion Criteria:

* children and young adults (between 2 to 25 years old)

Exclusion Criteria:

* children below 2 years old
* adults more than 25 years old

Ages: 2 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Study population will be chosen by random sampling technique among children and young adults (between 2 to 25 years old) attending internal medicine and pediatric out- patient clinics at Sohag University hospital.
Sampling Method: Probability Sample
Enrollment: 667 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Studying prevalence of Helicobacter Pylori infection in children and young adults in Sohag governorate | 12 weeks following the startpoint of the study.
  determine the prevalence of Helicobacter Pylori infection in children and young adults in Sohag governorate by examining stool samples from 667 patients to detect h.pylori antigen

SECONDARY OUTCOMES:
detecting risk factors related to Helicobacter Pylori infection in children and young adults in sohag governorate | 12 weeks following the startpoint of the study
  We will use a semi-structured questionnaire to detect helicobacter pylori risk factors which include the following : Socio-demographic data, personal habits, physical activity and exercises, history of symptoms suggesting helicopter pylori infection like episodes of epigastric pain, vomiting and dyspepsia and family history, medication and comorbidities .

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine-Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided